CLINICAL TRIAL: NCT03110523
Title: A Phase 3, Multicenter, 22-Week, Double-Blind and 30-Week Open-Label Study to Evaluate the Efficacy and Safety of X0002 Spray in Relief of the Signs and Symptoms of Subjects With Osteoarthritis of the Lumbar Spine
Brief Title: A Study to Evaluate the Efficacy and Safety of X0002 Spray in Subjects With Osteoarthritis of the Lumbar Spine
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic business decision
Sponsor: Techfields Pharma Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TF-X0002-32
Record Dates: First submitted 2017-03-10; First posted 2017-04-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Osteoarthritis of the Lumbar Spine; Pain, Back
Keywords: Osteoarthritis, Lumbar Spine; Pain
MeSH Terms: conditions — Osteoarthritis, Spine; Back Pain; Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): High Dose: X0002 or placebo, BID (in the morning and before going to bed), n=376
  Interventions: Drug: X0002
- Group B (Experimental): Low Dose: X0002 or placebo, BID (in the morning and before going to bed), n=376
  Interventions: Drug: X0002

INTERVENTIONS:
Drug: X0002 — All subjects who provide informed consent will initiate the Screening Period of at least 14 (±3) days for the assessment of eligibility including radiographic evaluation of the lumbar spine. X-ray images must be collected within 4-11 hours after the subject wakes up. Those subjects who meet preliminary eligibility criteria will be treated with placebo in a subject-blind manner for 14(±3) days from Screening Visit to Day 1. Subjects with a placebo response exceeding 25% improvement in the average NPRS score over the previous 7 days will be excluded. Subjects with a Lane grading of 1 or 2 on their neutral lateral lumbar spine film per the central radiologist are eligible to be enrolled. At Day 1, eligible subjects will be randomly assigned to 1 of 2 treatment groups in a 1:1 ratio with a 1:1 ratio of active:placebo within each treatment group, and stratified evenly according to Lane Radiographic Grading Scale summary score (1 or 2) and gender.
  Other Names: X-0002

SUMMARY:
This is a Phase 3, Multicenter, Randomized, 22 Week, Double-Blind, Placebo Controlled and 3-Week, Open-Label Study to Evaluate the Efficacy and Safety of X0002 Spray in relief of the signs and symptoms of Subjects with Osteoarthritis of the Lumbar Spine. To evaluate the efficacy of X0002 spray compared to placebo for the relief of low back pain disability in subjects with osteoarthritis (OA) of the low back.

DETAILED DESCRIPTION:
All subjects who provide informed consent will initiate the Screening Period of at least 14 (±3) days for the assessment of eligibility including radiographic evaluation of the lumbar spine. X-ray images must be collected within 4-11 hours after the subject wakes up. Those subjects who meet preliminary eligibility criteria will be treated with placebo in a subject-blind manner for 14(±3) days from Screening Visit to Day 1. Subjects with a placebo response exceeding 25% improvement in the average Numeric Pain Rating Scale (NPRS) score over the previous 7 days will be excluded. Subjects with a Lane grading of 1 or 2 on their neutral lateral lumbar spine film per the central radiologist are eligible to be enrolled. At Baseline (Day 1), eligible subjects will be randomly assigned to 1 of 2 treatment groups in a 1:1 ratio with a 1:1 ratio of active:placebo within each treatment group (i.e., 1 subject to active treatment and 1 subject to placebo), and stratified evenly according to Lane Radiographic Grading Scale summary score (1 or 2) and gender.

Low back pain intensity as assessed by the average of the NPRS scores recorded in the eDiary for the 7 days prior to the visit will be used for the primary efficacy endpoint as well as secondary efficacy endpoints. Efficacy assessments will be conducted at Screening, and at visits at Day 1 (Baseline) Week 2, Week 4, Week 8, Week 12, Week 22, Week 32, Week 42, and Week 52 (EOT). The patient reported outcomes of Oswestry Disability Index (ODI), Subject Global Assessment, modified Brief Pain Inventory (mBPI) Severity score, mBPI Interference Score, Subject's Clinical Global Impression of Improvement (CGI-I), and Short Form 36-item Health Survey (SF-36) will be used for the secondary or exploratory efficacy endpoints.

Safety assessments will be performed at each scheduled visit and will include assessment of AEs, vital signs (blood pressure, pulse rate, respiratory rate, and oral temperature), clinical laboratories, physical examination, skin irritation, and electrocardiograms (ECGs) as indicated in the schedule of events. Phone calls will be made to the subject by a qualified staff member at the site every 2 weeks between scheduled visits where applicable to collect additional information related to AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to read and to provide written, personally signed, and dated informed consent to participate in the study, in accordance with the ICH GCP Guideline E6 and applicable regulations, before completing any study related procedures.
2. Has an understanding, ability, and willingness to fully comply with study procedures and restrictions, as determined by the investigator.
3. Must be a male or female between 35 and 85 years of age, inclusive.
4. Must have a body mass index between 18.5 and 40.0 kg/m2, inclusive.
5. Must have a history (documented diagnosis) of clinically symptomatic OA of the lumbar spine for ≥3 months at Screening.
6. Must have a Lane Radiographic Grading Scale summary score for lumbar spine OA (levels L1 through L5) of 1 or 2 as determined by a central radiologist at Screening.
7. Must have had low back pain while standing, walking, and/or on motion for at least 14 days during the month prior to Screening per subject self-report documented by the investigator.
8. Must have a score ≥4 and ≤9 on a 0 to 10 (11 point) NPRS (without analgesic medication other than rescue medication provided by the Sponsor) over the previous 7 days prior to Baseline (Day 1).
9. Must have an ODI score ≥40% and ≤90 % at Screening Visit and Baseline (Day 1).
10. With the exception of OA of the lumbar spine, must be in good general health with no clinically significant findings from medical history, vital signs, physical examination, ECG, and routine laboratory tests that could interfere with subject safety, pain or functional assessments, as determined by the investigator.
11. Female subjects must either not be of childbearing potential defined as 1) postmenopausal for at least 1 year; follicle stimulating hormone [FSH] must be in postmenopausal range for the central lab if used to confirm postmenopausal status in a woman not using estrogen replacement therapy OR 2) surgically sterile [i.e., bilateral tubal ligation, bilateral oophorectomy, or hysterectomy]) or be willing to practice abstinence or at least 1 of the following medically acceptable methods of birth control:

    * Hormonal methods such as oral, implantable, injectable, vaginal ring, or transdermal contraceptives for a minimum of 1 full cycle (based on the subject's usual menstrual cycle period) before study drug administration;
    * Intrauterine device;
    * Double-barrier method (condoms, sponge, or diaphragm with spermicidal jellies or cream).

Exclusion Criteria:

1. 1. Not willing to avoid unaccustomed, strenuous physical activity (e.g., starting a new weight lifting routine) for the duration of the study starting at Screening Visit and through their completion of participation in the study. Normal physical activity is allowed.
2. Has an active or pending workman's compensation claim or litigation related to back pain.
3. Has secondary OA of the low back or OA of lower limb joints that, in the opinion of the investigator, could interfere with pain and functional assessments related to the low back.
4. Has a history of spinal surgery.
5. Has more than 25% improvement from Numeric Pain Rating Scale (NPRS) score at the Screening visit to the average NPRS score over the previous 7 days prior to Day 1.
6. Has had significant injury, as judged by the investigator, involving the back within the 6 months before Screening.
7. Has been diagnosed with or has signs and symptoms of a radiculopathy, e.g., numbness or tingling in a dermatomal distribution of a lower limb, sciatica, as well as etiologies of low back pain other than OA.
8. Has skin lesions or wounds on or near the lumbar spine area to be treated at Screening or on Day 1, which may influence absorption of the medication or confound safety assessments per the investigator's opinion.
9. Has used gabapentin, pregabalin, antiepileptics, or specific antidepressants (i.e., tricyclics, serotonin norepinephrine reuptake inhibitors, or selective serotonin reuptake inhibitors) to treat pain in the 14 days before Screening. Other uses not related to the pain treatment may be permitted at the medical monitor's discretion provided they have been at a stable dose for at least 90 days.
10. Has had injections of corticosteroids, botulinum toxin, or viscosupplements (e.g., Synvisc®) to the spine area (eg., intra articular [IA], epidural or paraspinal) within the 12 weeks before Screening.
11. Has had IA, intradiscal or intravenous (IV) stem cell therapy in the 6 months prior to Screening.
12. Has received concomitant non-pharmacologic treatments (e.g., physiotherapy, acupuncture) that per investigator opinion could confound efficacy assessments within 14 days of Day 1.
13. Is not willing to discontinue any NSAIDs or other analgesics (i.e., acetaminophen other than rescue medication supplied by the Sponsor, and cyclooxygenase-2 [COX-2] inhibitors), other treatments such as cannabis, and any topical therapies (e.g., anesthetics, capsaicin) or potentially confounding concomitant nonpharmacologic treatments (e.g., physiotherapy, acupuncture) starting at Screening Visit until completing participation in the study (the use of ≤325 mg acetylsalicylic acid per day for cardiac prophylaxis is permitted).
14. Is not willing to discontinue applying any topical preparations containing Vitamin A acids (including all trans retinoic acid [tretinoin], 13 cis retinoic acid [isotretinoin], 9 cis retinoic acid [alitretinoin], Vitamin A [retinol], retinal, and their derivatives) to the low back starting at Screening Visit until completing participation in the study. Topical preparations containing Vitamin A acids or retinol may be applied to areas of the skin above the shoulders or to the lower extremities.
15. Has a history of significant hypersensitivity, intolerance, or allergy to ibuprofen, any other NSAIDs, aspirin, or acetaminophen.
16. Has used an anticoagulant or antiplatelet agent (except aspirin up to 325 mg/day for cardiac prophylaxis) in the 30 days prior to Screening.
17. Has had an active gastrointestinal (GI) ulceration in the 6 months prior to Screening or a history of GI bleeding within 5 years of Screening.
18. Has uncontrolled depression or other uncontrolled psychiatric disorder (subjects with controlled depression or other psychiatric disorder, if using medication, must be on a stable dose of a medication other than an epileptic, tricyclic, serotonin norepinephrine reuptake inhibitor, or selective reuptake inhibitor for ≥12 weeks prior to Screening to participate in the study).
19. Has positive results on fecal occult blood testing at Screening or on Day 1.
20. Has a documented history of chronic inflammatory disease (such as rheumatoid arthritis, ankylosing spondylitis, axial spondyloarthropathy, psoriatic arthritis, inflammatory bowel disease or gouty arthritis) or a chronic pain condition (such as fibromyalgia), or has other conditions that may affect the spine or the functional and pain assessments (e.g., diffuse idiopathic skeletal hyperostosis, spinal stenosis, osteoporosis, severe scoliosis [curvature >30 degrees], severe kyphosis or lordosis [curvature >50 degrees]).
21. Is an asthmatic requiring treatment with systemic corticosteroids in the last year. Asthmatic subjects using inhaled corticosteroids are eligible.
22. Has uncontrolled hypertension defined as systolic blood pressure >170 mmHg or diastolic blood pressure >90 mmHg at Baseline (may be repeated 1 additional time after 5 minutes rest to verify). The investigator may, at his discretion, choose to exclude subjects with blood pressure levels lower than these if he deems it in the best interest of the subject.
23. Is receiving systemic chemotherapy, has an active malignancy, lymphoproliferative disorder or blood dyscrasia of any type, or has been diagnosed with cancer within 5 years before Screening. Subjects with completely excised and healed squamous or basal cell carcinoma of the skin will be allowed.
24. Has had any osteoporosis treatments (e.g., bisphosphonates, denosumab, parathyroid hormone (PTH), strontium ranelate).
25. Has any other clinically significant unstable cardiovascular, respiratory, neurological, immunological, hematological, hepatic or renal disease, or any other condition that, in the investigator's opinion, could compromise the subject's welfare, ability to communicate with the study staff, or otherwise contraindicate study participation.
26. Has an abnormal clinical central laboratory assessment at Screening for any of the following:

    * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase or lactate dehydrogenase (LDH) ≥3 × the upper limit of normal [ULN]
    * Total bilirubin ≥1.5 × ULN
    * Creatinine ≥1.5 × ULN
    * Hemoglobin <10 g/dL
27. Has any other clinically significant central laboratory finding at Screening that in the investigator's opinion contraindicates study participation;
28. Has clinically significant abnormality on 12-lead ECG, including a QTcF interval >450 milliseconds for males and 470 msec for females.
29. Is pregnant, planning to become pregnant during the study, or lactating; for women of childbearing potential, serum and urine pregnancy test must be negative at Screening Visit and urine pregnancy test must be negative at Baseline (Day 1) for subject to be eligible to participate.
30. Has participated in a previous clinical study with X0002.
31. Has participated in any other investigational clinical trial within the past 30 days or 5 half-lives of the investigational drug, whichever is longer, prior to Screening.
32. Has known alcohol or other substance abuse in the investigator's opinion.
33. Is a participating investigator, sub-investigator, study coordinator, or employee of a participating investigator, or is an immediate family member of the aforementioned.
34. Has any factor, which in the opinion of the investigator would jeopardize the evaluation or safety or be associated with poor adherence to the protocol.
35. Does not have access to telephone and/or ability to gain technology access.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Average daily Numeric Pain Rating Scale (NPRS) score [0 (no pain) to 10 (worst pain imaginable] for the 7 days prior to Week 12 | Week 12
  Change from Baseline in the average daily NPRS score for the 7 days prior to Week 12

SECONDARY OUTCOMES:
Average daily Numeric Pain Rating Scale (NPRS) score [0 (no pain) to 10 (worst pain imaginable] for the 7 days prior to Weeks 2, 4, 8, and 22 | Week 2, 4, 8, and 22
  Change from Baseline in the average daily NPRS score for the 7 days prior to Weeks 2, 4, 8, and 22
Oswestry Disability Index (ODI) score ( 0 is equated with no disability and 100 is the maximum disability possible) at Weeks 2, 4, 8, 12, and 22 | Week 2, 4, 8, 12, and 22
  Change from Baseline in the ODI score at Weeks 2, 4, 8, 12, and 22
Subject Global Assessment of disease status at Weeks 2, 4, 8, 12, and 22 | Week 2, 4, 8, 12, and 22
  To evaluate the effect of X0002 spray for change of Subject Global Assessment of disease status in subjects with OA of the lumbar spine
Modified Brief Pain Inventory (mBPI)-Severity score (on a scale ranging from 0 to 10; '0=No pain and 10=Pain as bad as you can imagine) at Weeks 2, 4, 8, 12, and 22 | Week 2, 4, 8, 12, and 22
  To evaluate the change from Baseline in the mBPI-Severity score at Weeks 2, 4, 8, 12, and 22
Modified Brief Pain Inventory (mBPI)-Interference score (on a scale ranging from 0 to 10 assessing how pain has interfered with certain functions in the previous 24 hours; '0=Does not interfere and 10=Completely interferes) at Weeks 2, 4, 8, 12, and 22 | Week 2, 4, 8, 12, and 22
  To evaluate the effect of X0002 spray for change mBPI-Severity score in subjects with OA of the lumbar spine.
Subject Clinician's Clinical Global Impression-Improvement (CGI-I) Score (1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse) at Weeks 2, 4, 8, 12, and 22 | Week 2, 4, 8, 12, and 22
  To evaluate the change from the Baseline in the Subject CGI-I at Weeks 2, 4, 8, 12, and 22
Average rescue medication (acetaminophen) consumed for low back pain at Weeks 2, 4, 8, 12, and 22. | Week 2, 4, 8, 12, and 22
  To evaluate the change of the average daily dose in mg of rescue medication (acetaminophen) consumed for low back pain at Weeks 2, 4, 8, 12, and 22.(acetaminophen) consumed for low back pain in subjects with OA of the lumbar spine between 2 visits.
Mental Component Summary (MCS) score (lower the score is the more disability) at Weeks 2, 4, 8, 12, and 22 | Week 2, 4, 8, 12, and 22
  To evaluate the change from Baseline in the SF-36v2 overall score, Physical Component Summary (PCS) score, and Mental Component Summary (MCS) score at Weeks 2, 4, 8, 12, and 22.

IPD SHARING:
Plan to Share IPD: No